CLINICAL TRIAL: NCT06206954
Title: Increasing Initiation of Evidence-based Weight Loss Treatment
Brief Title: Supporting Decisions on Lifestyle Change
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB202300516; R01DK134409 (NIH)
Record Dates: First submitted 2024-01-02; First posted 2024-01-16 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Obesity
Keywords: initiation; recruitment; engagement; behavioral intervention
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Parallel cluster randomized
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators (with exception of statistician) will be masked to study condition. Outcome assessors and all staff engaging directly with participants will be masked to study condition, except those staff who are sending intervention content.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MyHealthPath Tool (Experimental): Receive MyHealthPath Tool intervention.
  Interventions: Behavioral: MyHealthPath Tool
- MyHealthPath Guide (Active Comparator): Receive MyHealthPath Guide intervention
  Interventions: Behavioral: MyHealthPath Guide

INTERVENTIONS:
Behavioral: MyHealthPath Tool — Tailored, brief online tool to help patients learn about weight treatment options
  Arms: MyHealthPath Tool
Behavioral: MyHealthPath Guide — Informational material to help patients learn about weight treatment options
  Arms: MyHealthPath Guide

SUMMARY:
This study will test the effects of a brief, individually tailored intervention aiming to increase initiation of comprehensive behavioral weight loss treatment on weight.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Body Mass Index (BMI) ≥ 30 kg/m2 based on self-report body weight and height, or BMI ≥ 27-29.9 kg/m2 with a weight related comorbidity of hypertension, type 2 diabetes, pre-diabetes, dyslipidemia, or obstructive sleep apnea, gastroesophageal reflux disease, or coronary artery disease.
* Self-report weight ≤ 375 lbs (the maximum weight that BodyTrace scales can accurately detect is 397 lbs, thus 375 lbs provides a buffer to allow detection of at least 20 lbs weight gain).
* Has a desire to weigh less
* Has valid email address in Electronic Health Record
* Has an appointment scheduled with enrolled PCP about 21-28 days after electronic data pull
* Speaks and reads English
* Has either WiFi internet access at home or a phone or tablet with a data plan.

Exclusion criteria

* Currently enrolled in evidence-based comprehensive weight loss treatment
* Pregnant or planning to become pregnant in the next 6 months
* Currently breastfeeding (or pumping breastmilk) more than 3 times per day.
* Currently undergoing treatment for cancer
* Had cardiovascular event in the past 60 days
* Severe depression symptoms on PHQ-8 (total score ≥20)
* Inpatient psychiatric treatment in the past 6 months
* Eating disorder in past 5 years
* Congestive heart failure resulting in recent (past 6 months) hospitalization or contributing to difficulty breathing or difficulty doing daily activities.
* Dementia diagnosis
* Bariatric surgery in the past year or currently undergoing evaluation for bariatric surgery
* Currently taking doctor-prescribed medication for weight loss
* Inability to stand on body weight scale independently
* Impaired hearing
* Unable to read content on websites without assistance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Proportion initiating treatment | Within 2 months of PCP appointment date
  Attend at least one intervention session of comprehensive behavioral weight loss intervention. Documented by interventionist/program.

SECONDARY OUTCOMES:
Number of treatment sessions attended | 6 months
  Total number of attended intervention session of comprehensive behavioral weight loss intervention. Documented by interventionist/program.
Proportion discussing weight-related topic with PCP | at completion of PCP visit (occuring up to 4 weeks after enrollment)
  Per patient self-report, discussed weight, diet, or physical activity with PCP at index PCP visit.
Proportion achieving 5% weight loss | 6 months
  Proportion of participants losing 5% of their baseline weight between baseline and 6 months
Percent weight loss | 6 months
  Percent weight loss from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Megan A McVay, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data will be shared with other researchers. Researchers may need to complete a data use authorization agreement.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available within one year of study completion and remain available indefinitely.
Access Criteria: Access will be granted to researchers for any scientific purpose, including verifying/replicating analyses or conducting additional analyses, or